CLINICAL TRIAL: NCT00322556
Title: A Multicenter Extension Study on the Safety and Efficacy of IgPro10 in Patients With Primary Immunodeficiency (PID)
Brief Title: Safety and Efficacy of Intravenous Immunoglobulin IgPro10 in Patients With Primary Immunodeficiencies (PID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLB05_006CR
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-09

CONDITIONS: Agammaglobulinemia; IgG Deficiency; Common Variable Immunodeficiency
Keywords: Immunoglobulin Intravenous; Agammaglobulinemia; Hypogammaglobulinemia; Common variable immunodeficiency; Immunoglobulin G; Children
MeSH Terms: conditions — Agammaglobulinemia; IgG Deficiency; Common Variable Immunodeficiency | interventions — Immunoglobulins, Intravenous

ARMS (1):
- IgPro10 (Experimental): See Intervention Description
  Interventions: Drug: Immunoglobulins Intravenous (Human)

INTERVENTIONS:
Drug: Immunoglobulins Intravenous (Human) — Liquid formulation; treatment schedule every 3 or 4 weeks using an individualized regimen with a dose of 0.2 - 0.8 g IgG per kg bw

SUMMARY:
The objectives of this trial are the assessment of safety and efficacy of IgPro10 in patients with PID, and the assessment of tolerability of high infusion rates. To demonstrate safety, the number of infusions temporally associated with AEs, the rate, severity and relationship of all AEs and the vital sign changes during each infusion will be evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

Patients with CVID (Common Variable Immunodeficiency) or XLA (X-linked agammaglobulinemia) who:

Participated in the Phase III clinical study with intravenous IgPro10 (study number ZLB03_002CR) at 3- or 4- weekly intervals for 12 months (referred to as 'old' subjects)

OR

Were ≥ 6 years of age, were on other stable intravenous immunoglobulin therapy (200-800 mg IgG per kg body weight) at 3- or 4-week intervals for at least 6 months, AND were interested in participating in the Phase III clinical study with subcutaneous IgPro20 (study number ZLB04_009CR) (referred to as 'new' subjects)

Written informed consent

Key Exclusion Criteria:

Diagnosis of epilepsia

Insulin dependent diabetes

Administration of steroids (daily ≥ 0.15 mg prednisone equivalent/kg/day) or other immunosuppressive drugs

History of cardiac insufficiency (NYHA III/IV), cardiomyopathy, congestive heart failure, severe hypertension

Ages: 4 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Coordinator, Study Director — CSL Behring
Locations (10):
- United States (10):
  - Contact CSL Behring for facility details, Los Angeles, California
  - Contact CSL Behring for facility details, Centennial, Colorado
  - Contact CSL Behring for facility details, North Palm Beach, Florida
  - Contact CSL Behring for facility details, St. Petersburg, Florida
  - Contact CSL Behring for facility details, Fort Wayne, Indiana
  - Contact CSL Behring for facility details, Indianapolis, Indiana
  - Contact CSL Behring for facility details, Iowa City, Iowa
  - Contact CSL Behring for facility details, Rochester, Minnesota
  - Contact CSL Behring for facility details, St Louis, Missouri
  - Contact CSL Behring for facility details, Dallas, Texas

REFERENCES:
- [Result] Sleasman JW, Duff CM, Dunaway T, Rojavin MA, Stein MR. Tolerability of a new 10% liquid immunoglobulin for intravenous use, Privigen, at different infusion rates. J Clin Immunol. 2010 May;30(3):442-8. doi: 10.1007/s10875-010-9373-x. Epub 2010 Mar 10. PMID 20217199

RESULTS

PARTICIPANT FLOW:
Groups:
- IgPro10: A 10% liquid formulation of human immunoglobulin G (stabilized with 250 millimole per liter of L-proline) administered as an intravenous infusion, every 3 or 4 weeks for the duration of the study.
Period: Overall Study
Arm/Group | IgPro10
Started | 55
Completed | 43
Not Completed | 12
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 3
Not completed — Other Reason | 7

BASELINE CHARACTERISTICS:
Arm/Group | IgPro10
Number analyzed (Participants) | 55
Age Continuous [Mean (Standard Deviation); unit: years] | 30 (21)
Age, Customized [Number; unit: participants]
  3 to < 12 years | 13
  12 to < 16 years | 8
  16 to < 65 years | 30
  >= 65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Infusions With One or More Temporally-associated Adverse Events (AEs).
Description: AEs were considered temporally-associated AEs if they occurred during the infusion or in the period from the start of the infusion until either 48 or 72 hours after the end of the infusion.
Time Frame: During each infusion, and within 48 or 72 hours after the end of each infusion.
Population: The Safety Data Set (SDS) comprised all subjects treated with the study drug.
Measure: Number; unit: Proportion of infusions
Units Other Than Participants: Infusions
Arm/Group | IgPro10
Number analyzed (Participants) | 55
Number analyzed (Infusions) | 771
Proportion of infusions
  During infusion | 0.073
  Within 48 hours after infusion | 0.141
  Within 72 hours after infusion | 0.150

2. Primary Outcome: Influence of Infusion Rate on Temporally-Associated AEs
Description: The total and most frequent (1% or more) number of infusions for which subjects experienced temporally-associated AEs occurring within 72 hours of infusion, by infusion rate (≤ 4 mg/kg/min, ≤ 8 mg/kg/min, and > 8 and ≤ 12 mg/kg/min).
  AEs were considered to be temporally-associated AEs if they occurred in the period from the start of the infusion until 72 hours after the end of the infusion.
Time Frame: Within 72 hours after each infusion
Population: 'New subjects' could receive IgPro10 at up to 4 mg/kg/min. 'Old' subjects (ie, those treated with the study drug who participated in a preceding, pivotal, Phase III clinical study with intravenous IgPro10 [study number ZLB03_002CR, NCT00168025]), could receive IgPro10 at up to 12 mg/kg/min at the discretion of the Investigator.
Measure: Number; unit: Infusions
Units Other Than Participants: Infusions
Groups:
- IgPro10 (≤ 4 mg/kg/Min): A 10% liquid formulation of human immunoglobulin G (stabilized with 250 millimole per liter of L-proline) administered as an intravenous infusion, every 3 or 4 weeks for the duration of the study, at the maximum infusion rate (≤ 4 mg/kg/min) for new subjects.
- IgPro10 (≤ 8 mg/kg/Min): A 10% liquid formulation of human immunoglobulin G (stabilized with 250 millimole per liter of L-proline) administered as an intravenous infusion, every 3 or 4 weeks for the duration of the study, at the low maximum infusion rate (≤ 8 mg/kg/min) for old subjects.
- IgPro10 (> 8 to ≤ 12 mg/kg/Min): A 10% liquid formulation of human immunoglobulin G (stabilized with 250 millimole per liter of L-proline) administered as an intravenous infusion, every 3 or 4 weeks for the duration of the study, at the high maximum infusion rate (> 8 and ≤ 12 mg/kg/min) for old subjects.
Arm/Group | IgPro10 (≤ 4 mg/kg/Min) | IgPro10 (≤ 8 mg/kg/Min) | IgPro10 (> 8 to ≤ 12 mg/kg/Min)
Number analyzed (Participants) | 10 | 22 | 23
Number analyzed (Infusions) | 81 | 423 | 265
Infusions
  All temporally-associated AEs | 23 | 153 | 30
  Headache | 10 | 54 | 2
  Pyrexia | 0 | 9 | 1
  Nausea | 0 | 8 | 2
  Back pain | 0 | 8 | 0
  Chills | 0 | 7 | 0
  Pain | 0 | 6 | 0
  Anaemia | 1 | 0 | 0
  Constipation | 2 | 0 | 0
  Fatigue | 3 | 0 | 0
  Influenza like illness | 3 | 1 | 0
  Myalgia | 1 | 0 | 0
  Pharyngolaryngeal pain | 1 | 1 | 2
  Eczema | 1 | 0 | 0
  Night sweats | 1 | 0 | 0

3. Primary Outcome: Rate of AEs by Severity and Relationship
Description: The AE rate was the number of AEs over the number of infusions administered.
  Mild AEs: Did not interfere with daily activities; Moderate AEs: Interfered with routine daily activities; Severe AEs: Impossible to perform routine daily activities.
  At least possibly related AEs included possibly related AEs, probably related AEs, and related AEs.
Time Frame: For the duration of the study, up to approximately 29 months
Population: The SDS comprised all subjects treated with the study drug.
Measure: Number; unit: AEs per infusion
Units Other Than Participants: infusions
Arm/Group | IgPro10
Number analyzed (Participants) | 55
Number analyzed (infusions) | 771
AEs per infusion
  All mild AEs | 0.467
  All moderate AEs | 0.280
  All severe AEs | 0.058
  Unrelated AEs | 0.610
  Possibly related AEs | 0.088
  Probably related AEs | 0.048
  Related AEs | 0.060
  At least possibly related mild AEs | 0.121
  At least possibly related moderate AEs | 0.062
  At least possibly related severe AEs | 0.013
  Unrelated mild AEs | 0.346
  Unrelated moderate AEs | 0.218
  Unrelated severe AEs | 0.045

4. Secondary Outcome: Annualized Rate of Acute Serious Bacterial Infections.
Description: The annualized rate was based on the total number of infections and the total number of subject study days for all subjects in the specified analysis population and adjusted to 365 days.
  Acute serious bacterial infections included pneumonia, bacteremia / septicemia, osteomyelitis / septic arthritis, bacterial meningitis, and visceral abscess.
Time Frame: For the duration of the study, up to approximately 29 months
Population: The Intention-To-Treat (ITT) data set comprised all subjects treated with the study drug
Measure: Number; unit: Infections per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro10
Number analyzed (Participants) | 55
Number analyzed (Subject Study Days) | 20757
Infections per subject year | 0.018

5. Secondary Outcome: Number of Days Out of Work / School / Kindergarten / Day Care or Inability to Perform Normal Activities Due to Illness.
Time Frame: For the duration of the study, up to approximately 29 months.
Population: The ITT data set comprised all subjects treated with the study drug. The patient diary (in which the number of days was recorded) was not available for 1 subject so the analyzed population was reduced from 55 to 54 subjects for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | IgPro10
Number analyzed (Participants) | 54
Days | 8.5 [0.0 to 104.0]

6. Secondary Outcome: Number of Days of Hospitalization.
Time Frame: For the duration of the study, up to approximately 29 months
Population: as for outcome 5
Measure: Median (Full Range); unit: Days
Arm/Group | IgPro10
Number analyzed (Participants) | 54
Days | 0.0 [0.0 to 17.0]

7. Secondary Outcome: Annualized Rate of Any Infection.
Description: The annualized rate was based on the total number of infections and the total number of subject study days for all subjects in the specified analysis population and adjusted to 365 days.
  Infections were classified as all AEs with the system organ class "infections and infestations" and AEs with the preferred term "conjunctivitis".
Time Frame: For the duration of the study, up to approximately 29 months.
Population: The ITT data set comprised all subjects treated with the study drug.
Measure: Number; unit: Infections per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro10
Number analyzed (Participants) | 55
Number analyzed (Subject Study Days) | 20757
Infections per subject year | 1.600

8. Secondary Outcome: Trough Levels of Total Immunoglobulin (IgG) Serum Concentrations.
Description: Mean IgG trough concentration. For this analysis, each subject's values were first aggregated to their median and the median values were then analyzed.
Time Frame: Prior to each infusion; every 3 or 4 weeks depending upon the dosing schedule.
Population: The ITT data set comprised all subjects treated with the study drug for which serum IgG information was available.
Measure: Mean (Full Range); unit: g/L
Arm/Group | IgPro10
Number analyzed (Participants) | 54
g/L | 9.72 [5.72 to 18.01]

9. Primary Outcome: Number of Subjects With Clinically Significant Changes in Vital Signs.
Description: Vital signs included heart rate, systolic blood pressure, diastolic blood pressure, and body temperature.
Time Frame: Before, during, and after each infusion.
Population: The Safety Data Set (SDS) comprised all subjects treated with the study drug.
Measure: Number; unit: Participants
Arm/Group | IgPro10
Number analyzed (Participants) | 55
Participants | 0

ADVERSE EVENTS:
Time Frame: For the duration of the study, up to approximately 29 months
Description: Only AEs starting at or after the first study drug infusion were included. The SDS comprised all subjects treated with the study drug.
Arm/Group | IgPro10
Serious Adverse Events (participants affected / at risk) | 11/55
Other Adverse Events (participants affected / at risk) | 48/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro10 (N=55)
Clostridial infection (Infections and infestations) | 1 (1)
Ileostomy closure (Surgical and medical procedures) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Giardiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Otitis externa fungal (Infections and infestations) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro10 (N=55)
Headache (Nervous system disorders) | 21 (147)
Sinusitis (Infections and infestations) | 14 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (17)
Nausea (Gastrointestinal disorders) | 11 (16)
Diarrhea (Gastrointestinal disorders) | 10 (13)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Pyrexia (General disorders) | 8 (22)
Vomiting (Gastrointestinal disorders) | 8 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (12)
Eczema (Skin and subcutaneous tissue disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Fatigue (General disorders) | 5 (9)
Nasopharyngitis (Infections and infestations) | 5 (5)
Pain (General disorders) | 5 (10)
Dizziness (Nervous system disorders) | 4 (4)
Hypertension (Vascular disorders) | 4 (6)
Insomnia (Psychiatric disorders) | 4 (4)
Pneumonia (Infections and infestations) | 3 (3)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Bronchitis (Infections and infestations) | 3 (3)
Chest pain (General disorders) | 3 (4)
Chills (General disorders) | 3 (7)
Conjunctivitis (Eye disorders) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 3 (4)
Gastroenteritis viral (Infections and infestations) | 3 (5)
Influenza-like illness (General disorders) | 3 (9)
Joint sprain (Injury, poisoning and procedural complications) | 3 (5)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Toothache (Gastrointestinal disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.